CLINICAL TRIAL: NCT01789970
Title: A 12-Week, Randomized, Double-Blind, Placebo-Controlled, Randomized-Withdrawal Study to Evaluate the Efficacy and Safety of Hydrocodone Bitartrate Extended-Release Tablets (CEP-33237) at 30 to 90 mg Every 12 Hours for Relief of Moderate to Severe Pain in Patients With Chronic Low Back Pain Who Require Opioid Treatment for an Extended Period of Time
Brief Title: Efficacy and Safety of Hydrocodone Bitartrate Extended-Release Tablets for Moderate to Severe Chronic Low Back Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C33237/3103
Record Dates: First submitted 2013-02-08; First posted 2013-02-12 (Estimated); Results first posted 2017-04-05 (Actual); Last update posted 2017-06-05 (Actual); Status verified 2017-06

CONDITIONS: Low Back Pain
Keywords: chronic low back pain; hydrocodone bitartrate; opioids
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Participants were administered hydrocodone ER tablets orally at dosages of 15, 30, 45, 60, or 90 mg every 12 hours at the dosage deemed successful for managing their pain during the titration period. During the treatment period, participants were administered placebo tablets twice a day that matched the dosage deemed successful for managing their pain during the titration period. A step-wise, double-blind schedule to tamper off active drug was implemented during the first 2 weeks of the 12-week, double-blind, placebo-controlled treatment period to reduce the risk of withdrawal effects in participants randomly assigned to placebo.
  Interventions: Drug: Hydrocodone ER; Drug: Placebo
- Hydrocodone ER (Experimental): Participants were administered hydrocodone ER tablets orally at dosages of 15, 30, 45, 60, or 90 mg every 12 hours at the dosage deemed successful for managing their pain during the titration period. During the 12-week, double-blind, placebo-controlled treatment period, participants randomly assigned to hydrocodone ER were administered tablets twice a day at the dosage deemed successful for managing their pain during the titration period.
  Interventions: Drug: Hydrocodone ER

INTERVENTIONS:
Drug: Hydrocodone ER — During the open-label, titration period, all participants were administered hydrocodone ER tablets at dosages of 15, 30, 45, 60, or 90 mg every 12 hours to identify a dosage deemed successful for managing their pain.
  Hydrocodone ER was taken by participants randomized to the hydrocodone ER treatment arm during the double-blind treatment period at the dose level identified during the titration period.
  Participants were instructed to take tablets with a glass of water on an empty stomach at least 1 hour before or 2 hours after eating.
  Other Names: CEP-33237; Hydrocodone bitartrate extended-release tablets
Drug: Placebo — Placebo matching the active drug dose identified during the titration period was taken by participants randomized to the placebo treatment arm during the double-blind treatment period.
  Participants were instructed to take intervention with a glass of water on an empty stomach at least 1 hour before or 2 hours after eating.
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate the efficacy of hydrocodone bitartrate extended-release tablets at doses of 30 to 90 mg every 12 hours compared with placebo in alleviating moderate to severe pain in patients with chronic low back pain. Patients may be opioid-naïve or opioid-experienced.

DETAILED DESCRIPTION:
The study consisted of a screening period of approximately 7 to 14 days, an open label titration period of up to 6 weeks, and a double blind treatment period of 12 weeks.

The objective of the open label titration period was to find the successful dose of hydrocodone extended release (ER) tablets that produced stable pain relief without unacceptable adverse events (AEs). Stable pain relief was defined as an average pain intensity (API) score over the previous 24 hours of 4 or less and a worst pain intensity (WPI) score of 6 or less on the 11-point numerical rating scale (NRS-11) (0=no pain to 10=worst pain imaginable) for either 4 consecutive days or 4 out of 7 consecutive days, while the same dose of study drug was maintained for up to 7 days. Scores for WPI and API were recorded daily in individual patient electronic diaries. Patients returned to the study center prior to each dose adjustment.

The starting dose of hydrocodone ER tablets depended on whether the subject was opioid-naïve or opioid-experienced. Opioid-naïve participants started at a 15-mg dose of hydrocodone ER tablets every 12 hours. For opioid-experienced participants, the starting dose of hydrocodone ER tablets was to be approximately equivalent to 50% of the dose of opioid analgesic that they were receiving at screening and administered every 12 hours. Investigators switched participants from previous opioid therapy to hydrocodone ER tablets on the basis of predefined dose equivalents.

Participants who met the criterion of a stabilized dose were randomly assigned into the 12 week, double-blind, placebo controlled treatment period on the final day of the open label titration period (baseline visit). Participants began treatment with double blind study drug at the effective dose of hydrocodone ER tablets achieved during the titration period or matching placebo. Rescue medication was permitted in addition to the study drug during the double blind treatment period.

Participants who participated in the study in compliance with the protocol and complete 12 weeks of double-blind treatment with study drug, were considered to have completed the study and could have been eligible to enroll in a 6-month open-label study (study C32337/3104, NCT01922739).

ELIGIBILITY:
Inclusion Criteria:

* The patient has had moderate to severe chronic low back pain for at least 3 months duration before screening.
* The patient is able to speak English and is willing to provide written informed consent, including a written opioid agreement, to participate in this study.
* The patient is willing and able to successfully self-administer the study drug, comply with study restrictions, complete the electronic diary, and return to the study center for scheduled study visits, as specified in the protocol.
* The patient is 18 through 80 years of age at the time of screening.
* Women of childbearing potential (not surgically sterile or 2 years postmenopausal) must use a medically accepted method of contraception, agree to continue use of this method for the duration of the study and for 30 days after participation in the study, and have a negative pregnancy test at screening. - Acceptable methods of contraception include barrier method with spermicide, intrauterine device (IUD), or steroidal contraceptive (oral, transdermal, implanted, and injected) in conjunction with a barrier method. NOTE: A woman will be considered surgically sterile if she has had a tubal ligation, hysterectomy, bilateral salpingo-oophorectomy or bilateral oophorectomy, or hysterectomy with bilateral salpingo-oophorectomy.
* Other criteria apply.

Exclusion Criteria:

* The patient is taking a total of more than 135 mg/day of oxycodone, or equivalent, during the 14 days before screening.
* The patient's primary painful condition under study is related to any source of chronic pain other than low back pain.
* The patient has radicular (nerve compression) pain or another type of purely neuropathic pain.
* The patient has known or suspected hypersensitivities, allergies, or other contraindications to any ingredient in the study drug.
* The patient has a recent history (within 5 years) or current evidence of alcohol or other substance abuse, with the exception of nicotine.
* The patient has medical or psychiatric disease that, in the opinion of the investigator, would compromise collected data.
* Other criteria apply.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 625 (Actual)
Dates: Start 2013-03; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Project Leader, Study Director — Teva GCO
Locations (87):
- United States (87):
  - Teva Investigational Site 10416, Anniston, Alabama
  - Teva Investigational Site 10382, Birmingham, Alabama
  - Teva Investigational Site 10403, Birmingham, Alabama
  - Teva Investigational Site 10412, Birmingham, Alabama
  - Teva Investigational Site 10426, Mobile, Alabama
  - Teva Investigational Site 10436, Montgomery, Alabama
  - Teva Investigational Site 10363, Phoenix, Arizona
  - Teva Investigational Site 10366, Phoenix, Arizona
  - Teva Investigational Site 10437, Tucson, Arizona
  - Teva Investigational Site 10358, Anaheim, California
  - Teva Investigational Site 10408, Bell Gardens, California
  - Teva Investigational Site 10425, Carmichael, California
  - Teva Investigational Site 10390, Cerritos, California
  - Teva Investigational Site 10429, El Cajon, California
  - Teva Investigational Site 10423, Escondido, California
  - Teva Investigational Site 10740, Garden Grove, California
  - Teva Investigational Site 10391, Huntington Park, California
  - Teva Investigational Site 10422, La Jolla, California
  - Teva Investigational Site 10413, Laguna Hills, California
  - Teva Investigational Site 10442, Laguna Hills, California
  - Teva Investigational Site 10370, Los Angeles, California
  - Teva Investigational Site 10392, Sherman Oaks, California
  - Teva Investigational Site 10398, Thousand Oaks, California
  - Teva Investigational Site 10428, Torrance, California
  - Teva Investigational Site 10361, Walnut Creek, California
  - Teva Investigational Site 10441, Waterbury, Connecticut
  - Teva Investigational Site 10369, DeLand, Florida
  - Teva Investigational Site 10744, Edgewater, Florida
  - Teva Investigational Site 10379, Fort Lauderdale, Florida
  - Teva Investigational Site 10365, Jacksonville, Florida
  - Teva Investigational Site 10445, Leesburg, Florida
  - Teva Investigational Site 10362, Orlando, Florida
  - Teva Investigational Site 10381, Ormond Beach, Florida
  - Teva Investigational Site 12036, Pembroke Pines, Florida
  - Teva Investigational Site 10357, Plantation, Florida
  - Teva Investigational Site 10367, Royal Palm Beach, Florida
  - Teva Investigational Site 10435, Royal Palm Beach, Florida
  - Teva Investigational Site 10742, Sanford, Florida
  - Teva Investigational Site 10432, Columbus, Georgia
  - Teva Investigational Site 10383, Marietta, Georgia
  - Teva Investigational Site 10385, Marietta, Georgia
  - Teva Investigational Site 10444, Newnan, Georgia
  - Teva Investigational Site 10431, Meridian, Idaho
  - Teva Investigational Site 10743, Meridian, Idaho
  - Teva Investigational Site 10411, Chicago, Illinois
  - Teva Investigational Site 10418, Avon, Indiana
  - Teva Investigational Site 10380, Evansville, Indiana
  - Teva Investigational Site 10440, Newburgh, Indiana
  - Teva Investigational Site 10375, Overland Park, Kansas
  - Teva Investigational Site 10419, New Orleans, Louisiana
  - Teva Investigational Site 10359, Shreveport, Louisiana
  - Teva Investigational Site 10389, Fall River, Massachusetts
  - Teva Investigational Site 10388, Bay City, Michigan
  - Teva Investigational Site 10397, Biloxi, Mississippi
  - Teva Investigational Site 10406, Hazelwood, Missouri
  - Teva Investigational Site 10401, St Louis, Missouri
  - Teva Investigational Site 10376, Omaha, Nebraska
  - Teva Investigational Site 10396, Omaha, Nebraska
  - Teva Investigational Site 10417, Henderson, Nevada
  - Teva Investigational Site 10399, Las Vegas, Nevada
  - Teva Investigational Site 10409, Berlin, New Jersey
  - Teva Investigational Site 10439, Buffalo, New York
  - Teva Investigational Site 10394, New York, New York
  - Teva Investigational Site 10407, New York, New York
  - Teva Investigational Site 10410, New York, New York
  - Teva Investigational Site 10443, Raleigh, North Carolina
  - Teva Investigational Site 10414, Winston-Salem, North Carolina
  - Teva Investigational Site 10446, Oklahoma City, Oklahoma
  - Teva Investigational Site 10415, Altoona, Pennsylvania
  - Teva Investigational Site 10430, Duncansville, Pennsylvania
  - Teva Investigational Site 10386, Mechanicsburg, Pennsylvania
  - Teva Investigational Site 10373, Tipton, Pennsylvania
  - Teva Investigational Site 10404, North Charleston, South Carolina
  - Teva Investigational Site 10741, Spartanburg, South Carolina
  - Teva Investigational Site 10405, Austin, Texas
  - Teva Investigational Site 10364, Dallas, Texas
  - Teva Investigational Site 10372, Dallas, Texas
  - Teva Investigational Site 10395, Dallas, Texas
  - Teva Investigational Site 10371, Houston, Texas
  - Teva Investigational Site 12035, Houston, Texas
  - Teva Investigational Site 10377, Lake Jackson, Texas
  - Teva Investigational Site 10374, Plano, Texas
  - Teva Investigational Site 10378, San Antonio, Texas
  - Teva Investigational Site 10402, Salt Lake City, Utah
  - Teva Investigational Site 10438, Roanoke, Virginia
  - Teva Investigational Site 10420, Bellevue, Washington
  - Teva Investigational Site 10433, Everett, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 845 patients with moderate to severe chronic low back pain were screened at 78 centers in the U.S.
Pre-assignment Details: Of the 625 patients enrolled, 2 patients withdrew consent before taking any study drug. Of 623 patients who were enrolled and received study drug, 371 patients achieved a successful dose of hydrocodone extended-release (ER) tablets and were randomly assigned to receive hydrocodone ER or placebo during the double-blind treatment period
Groups:
- Hydrocodone ER (Open-Label Titration Period): All participants were administered hydrocodone ER tablets at dosages of 15, 30, 45, 60, or 90 mg every 12 hours to identify a dosage deemed successful for managing their pain.
- Placebo (Double-blind Treatment Period): Participants were administered placebo tablets every 12 hours that matched the dosage deemed successful for managing their pain during the titration period. A step wise, double-blind tapering schedule was implemented during the first 2 weeks of the 12 week, double blind, placebo controlled treatment period to reduce the risk of withdrawal effects in patients randomly assigned to placebo.
- Hydrocodone ER (Double-blind Treatment Period): Participants were administered hydrocodone ER tablets at a dosage deemed successful for managing their pain during the titration period. Dosages of 15, 30, 45, 60, or 90 mg every 12 hours were given for 12 weeks during the double-blind period.
Period: Open-label Titration Period
Arm/Group | Hydrocodone ER (Open-Label Titration Period) | Placebo (Double-blind Treatment Period) | Hydrocodone ER (Double-blind Treatment Period)
Started | 625 | 0 | 0
Safety Analysis Set | 623 (Two enrolled patients were not treated) | 0 | 0
Completed | 371 | 0 | 0
Not Completed | 254 | 0 | 0
Not completed — Adverse Event | 68 | 0 | 0
Not completed — Lack of Efficacy | 31 | 0 | 0
Not completed — Withdrawal by Subject | 31 | 0 | 0
Not completed — Protocol Violation | 18 | 0 | 0
Not completed — Lost to Follow-up | 5 | 0 | 0
Not completed — Noncompliance to study drug admin | 11 | 0 | 0
Not completed — Noncompliance with study rescue meds | 2 | 0 | 0
Not completed — Noncompliance with study procedures | 8 | 0 | 0
Not completed — Pregnancy | 2 | 0 | 0
Not completed — Other | 76 | 0 | 0
Not completed — Dropped out prior to dosing | 2 | 0 | 0
Period: Double-blind Treatment Period (12 Weeks)
Arm/Group | Hydrocodone ER (Open-Label Titration Period) | Placebo (Double-blind Treatment Period) | Hydrocodone ER (Double-blind Treatment Period)
Started | 0 | 180 | 191
Full Analysis Set and Safety Set | 0 | 179 (One participant was randomized but not treated.) | 191
Completed | 0 | 130 | 147
Not Completed | 0 | 50 | 44
Not completed — Adverse Event | 0 | 9 | 15
Not completed — Lack of Efficacy | 0 | 17 | 5
Not completed — Withdrawal by Subject | 0 | 7 | 9
Not completed — Protocol Violation | 0 | 9 | 7
Not completed — Noncompliance to study drug admin | 0 | 2 | 2
Not completed — Noncompliance with study procedures | 0 | 2 | 1
Not completed — Lost to Follow-up | 0 | 1 | 2
Not completed — Pregnancy | 0 | 1 | 0
Not completed — Other | 0 | 1 | 3
Not completed — Dropped out prior to dosing | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent to treat population
Groups:
- Hydrocodone ER (Double-blind Treatment Period): Participants were administered extended-release hydrocodone tablets at a dosage deemed successful for managing their pain during the titration period. Dosages of 15, 30, 45, 60, or 90 mg every 12 hours were given for 12 weeks during the double-blind period.
- Total: Total of all reporting groups
Arm/Group | Placebo (Double-blind Treatment Period) | Hydrocodone ER (Double-blind Treatment Period) | Total
Number analyzed (Participants) | 180 | 191 | 371
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.8 (12.51) | 51.7 (13.48) | 51.8 (13.00)
Age, Customized [Count of Participants; unit: Participants]
  <= 65 years | 154 | 156 | 310
  > 65 years | 26 | 35 | 61
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92 | 97 | 189
  Male | 88 | 94 | 182
Race [Count of Participants; unit: Participants]
  White | 129 | 133 | 262
  Black | 41 | 39 | 80
  Asian | 8 | 13 | 21
  American Indian or Alaska Native | 2 | 2 | 4
  Native Hawaiian or other Pacific Islander | 0 | 1 | 1
  Other | 0 | 3 | 3
Ethnicity [Count of Participants; unit: Participants]
  Hispanic or Latino | 23 | 24 | 47
  Non-Hispanic and non-Latino | 156 | 167 | 323
  Unknown | 1 | 0 | 1
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 31.5 (8.22) | 31.3 (7.37) | 31.4 (7.78)
Participant Opioid Status [Count of Participants; unit: Participants] — Opioid-naïve patients were defined as those who were taking tramadol or less than 10 mg per day of oxycodone, or equivalent (including around-the-clock and rescue medication) for the 14 days before screening. Opioid-experienced patients were defined as those who were taking 10 mg or more per day of oxycodone, or equivalent (including around-the-clock and rescue medication) for the 14 days before screening. Opioid-experienced patients requiring more than 135 mg/day of oxycodone, or equivalent, during the 14 days before study entry were excluded from the study.
  Participants
    Opioid-naive | 105 | 110 | 215
    Opioid-experienced | 75 | 81 | 156
Duration Since Diagnosis of Chronic Low Back Pain [Mean (Standard Deviation); unit: years] | 11.5 (10.35) | 11.3 (10.29) | 11.4 (10.31)
Duration of Opioid Therapy [Mean (Standard Deviation); unit: years] | 2.9 (3.76) | 3.5 (4.85) | 3.2 (4.37)
Average Daily Hydrocodone Equivalent Dose [Mean (Standard Deviation); unit: mg] | 18.2 (28.55) | 22.1 (30.18) | 20.2 (29.43)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 12 of the Treatment Period in Weekly Average of Daily Worst Pain Intensity (WPI)
Description: The WPI was recorded daily by participants in an electronic diary using an 11-point numerical rating scale (NRS-11), a Likert-type scale in which 0=no pain and 10=the worst pain imaginable. Participants selected the number that best described their worst pain intensity over the last 24 hours. Weekly WPI scores averaged daily scores collected over the previous 7 days for each analysis visit. Negative change from baseline scores indicate improvement in pain control.
  The analysis included WPI data observed before discontinuation of study drug and was based on the multiple imputations (MI) method to handle missing scores at week 12. Consistent with the recommendations of the National Academy of Sciences (NAS) report (Panel on Handling Missing Data in Clinical Trials 2010), the MI method includes an assumption of missing at random (MAR) and takes into account a potential bias toward the active-drug treatment group for patients who discontinued study drug because of adverse events.
Time Frame: Days -6 to 0 of Treatment Period (baseline), Week 12 of Treatment Period
Population: The full analysis set, which includes all randomized participants who received at least 1 dose of study drug and had at least 1 post-baseline efficacy observation.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo (Double-blind Treatment Period) | Hydrocodone ER (Double-blind Treatment Period)
Number analyzed (Participants) | 179 | 191
units on a scale | 0.71 (0.145) | 0.07 (0.134)
Statistical Analysis 1: Comparison: Placebo (Double-blind Treatment Period) vs Hydrocodone ER (Double-blind Treatment Period); The least squares means of the change from baseline to week 12 in WPI were compared between the active drug and placebo treatment groups; Test type: Superiority or Other; p < 0.001, ANCOVA — 5% significance level; The model included treatment, study center, opioid status, and baseline WPI score; Mean Difference (Final Values) = 0.63, 95% CI 2-sided [0.26 to 1.00] — Placebo - Hydrocodone ER

2. Secondary Outcome: Change From Baseline to Week 12 of the Treatment Period in Weekly Average Pain Intensity (API)
Description: The API over the last 24 hours was recorded daily by patients in an electronic diary using an 11-point numerical rating scale (NRS-11), a Likert-type scale in which 0=no pain and 10=the worst pain imaginable. Participants selected the number that best described the average pain intensity over the last 24 hours. Weekly API scores averaged daily scores collected over the previous 7 days for each analysis visit. Negative change from baseline scores indicate improvement in pain control.
  The analysis included API data observed before discontinuation of study drug and was based on the MI method to handle missing scores at week 12. Consistent with the recommendations of the National Academy of Sciences (NAS) report (Panel on Handling Missing Data in Clinical Trials 2010), the MI method includes an assumption of missing at random (MAR) and takes into account a potential bias toward the active-drug treatment group for patients who discontinued study drug because of adverse events.
Time Frame: Days -6 to 0 of Treatment Period (baseline), Week 12
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo (Double-blind Treatment Period) | Hydrocodone ER (Double-blind Treatment Period)
Number analyzed (Participants) | 179 | 191
units on a scale | 0.57 (0.126) | 0.02 (0.116)
Statistical Analysis 1: Comparison: Placebo (Double-blind Treatment Period) vs Hydrocodone ER (Double-blind Treatment Period); The least squares means of the change from baseline to week 12 in API were compared between the active drug and placebo treatment groups; Test type: Superiority or Other; p < 0.001, ANCOVA — 5% significance level; The model included treatment, study center, opioid status, and baseline WPI score; Mean Difference (Final Values) = 0.58, 95% CI 2-sided [0.25 to 0.91] — Placebo - Hydrocodone ER

3. Secondary Outcome: Kaplan-Meier Estimates for Time to Loss of Efficacy
Description: Time to loss of efficacy was defined as discontinuation of study drug for lack of efficacy or the start of excessive rescue medication while taking study drug. Excessive rescue medication usage was defined as 10 or more days of rescue medication usage in any 14 consecutive days at a total of 15 mg (hydrocodone-equivalent) or higher each day during the post 2-week tapering period of the double-blind treatment period.
Time Frame: Day 1 to Week 12 of Treatment Period
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo (Double-blind Treatment Period) | Hydrocodone ER (Double-blind Treatment Period)
Number analyzed (Participants) | 179 | 191
days | NA [NA to NA] — Insufficient number of participants with loss of efficacy | NA [NA to NA] — Insufficient number of participants with loss of efficacy
Statistical Analysis 1: Comparison: Placebo (Double-blind Treatment Period) vs Hydrocodone ER (Double-blind Treatment Period); Test type: Superiority or Other; p = 0.059, Wald chi-square — 5% significance level; Cox proportional hazards model with treatment, baseline worst pain intensity (WPI), opioid status, and center in the model; Hazard Ratio (HR) = 0.68, 95% CI 2-sided [0.5 to 1.01]

4. Secondary Outcome: Percentage of Participants With a 30% or Greater Increase in Weekly Average Pain Intensity (API) From Baseline to Week 12 Visit, and an Average API Score of 5 or Higher at Week 12
Description: The API over the last 24 hours was recorded daily by participants in an electronic diary using an 11-point numerical rating scale (NRS-11), a Likert-type scale in which 0=no pain and 10=the worst pain imaginable. Participants selected the number that best described the average pain intensity over the last 24 hours. Weekly API scores averaged daily scores collected over the previous 7 days for each analysis visit.
Time Frame: Days -6 to 0 of Treatment Period (baseline), Week 12
Population: Full analysis set, including participants with observed weekly average API for week 12
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Double-blind Treatment Period) | Hydrocodone ER (Double-blind Treatment Period)
Number analyzed (Participants) | 133 | 152
percentage of participants
  API increase >=30% and API >=5 | 18.8 | 12.5
  API increase >=30% | 36.1 | 21.1
  API >=5 | 24.1 | 16.4
Statistical Analysis 1: Comparison: Placebo (Double-blind Treatment Period) vs Hydrocodone ER (Double-blind Treatment Period); API increase >=30% and API >=5; Test type: Superiority or Other; p = 0.0293, Regression, Logistic — 5% significance level; stratified by center with the following effects: treatment group, baseline API, and opioid status; Odds Ratio (OR) = 0.67, 95% CI 2-sided [0.47 to 0.96] — Hydrocodone ER / Placebo

5. Secondary Outcome: Change From Baseline to Final On-Treatment Visit in Roland Morris Disability Questionnaire (RMDQ) Score
Description: The RMDQ is a patient-rated, 24-question evaluation used to assess acute disability associated with low back pain. Each question is answered with a YES or NO response, and each YES response is given 1 point. Scores on the RMDQ range from 0 to 24, with higher scores indicating greater disability. Negative change from baseline scores indicate improvement in level of disability.
Time Frame: Days 7-14 of Titration Period (baseline), Week 12 or end of study visit during the Treatment Period
Population: Full analysis set, including participants with RMDQ score for the final on-treatment visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo (Double-blind Treatment Period) | Hydrocodone ER (Double-blind Treatment Period)
Number analyzed (Participants) | 171 | 178
units on a scale | -1.9 (4.47) | -1.5 (4.70)
Statistical Analysis 1: Comparison: Placebo (Double-blind Treatment Period) vs Hydrocodone ER (Double-blind Treatment Period); Test type: Superiority or Other; p = 0.557, ANCOVA — 5% significance level; Model with the following effects: treatment, study center, opioid status, and baseline RMDQ score; Mean Difference (Final Values) = -0.28, 95% CI 2-sided [-1.20 to 0.65] — Placebo - Hydrocodone ER

6. Secondary Outcome: Participants With Adverse Events During Open-Label Titration and Double-Blind Treatment Periods
Description: An adverse event (AE) was defined in the protocol as any untoward medical occurrence that develops or worsens in severity during the conduct of a clinical study and does not necessarily have a causal relationship to the study drug. Severity was rated by the investigator on a scale of mild, moderate and severe, with severe= an inability to carry out usual activities. Relation of AE to treatment was determined by the investigator. Serious AEs include death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, OR an important medical event that jeopardized the patient and required medical intervention to prevent the previously listed serious outcomes.
Time Frame: Day 1 of Titration Period up to Week 12 of Treatment Period (maximum treatment duration was 127 days)
Population: Safety analysis set (Titration Period) and Full analysis set (Treatment Period)
Measure: Count of Participants; unit: Participants
Groups:
- Opioid-Naive (Open-Label Titration Period): Opioid-naïve participants were defined as those who were taking tramadol or less than 10 mg per day of oxycodone, or equivalent (including around-the-clock and rescue medication) for the 14 days before screening.
  Opioid-naïve participants started at a 15-mg dose of hydrocodone ER tablets every 12 hours.
  All participants were administered hydrocodone ER tablets at dosages of 15, 30, 45, 60, or 90 mg every 12 hours to identify a dosage deemed successful for managing their pain.
- Opioid-Experienced (Open-Label Titration Period): Opioid-experienced participants were defined as those who were taking 10 mg or more per day of oxycodone, or equivalent (including around-the-clock and rescue medication) for the 14 days before screening.
  For opioid-experienced participants, the starting dose of hydrocodone ER tablets was to be approximately equivalent to 50% of the dose of opioid analgesic that they were receiving at screening and administered every 12 hours.
  All participants were administered hydrocodone ER tablets at dosages of 15, 30, 45, 60, or 90 mg every 12 hours to identify a dosage deemed successful for managing their pain.
Arm/Group | Opioid-Naive (Open-Label Titration Period) | Opioid-Experienced (Open-Label Titration Period) | Placebo (Double-blind Treatment Period) | Hydrocodone ER (Double-blind Treatment Period)
Number analyzed (Participants) | 368 | 255 | 179 | 191
Participants
  Any adverse event | 196 | 117 | 88 | 106
  Severe adverse event | 13 | 5 | 3 | 9
  Treatment-related adverse event | 166 | 81 | 50 | 67
  Deaths | 0 | 0 | 0 | 0
  Serious adverse event | 6 | 4 | 3 | 3
  Discontinued study drug treatment due to AE | 53 | 22 | 7 | 11

7. Secondary Outcome: Participants With Clinically Significant Hearing Changes From Baseline to Final Assessment in Pure Tone Audiometry Test Results
Description: Pure tone audiometry was performed by a qualified audiologist and was not done at the study center. During the test, the patient wore headphones and was seated in a quiet room; trained personnel manipulated the audiometry equipment to test the patient's hearing. For serial audiograms, the criteria for a clinically significant (CS) hearing change were based on the guidance from the American Speech-Language Hearing Association (ASHA) 1994 (Konrad-Martin et al 2005). These criteria included the following: greater than 20 decibels (dB) pure tone threshold shift at 1 frequency; greater than 10 dB shift at 2 consecutive test frequencies; or threshold response shifting to "no response" at 3 consecutive test frequencies.
Time Frame: Days 7-14 of Titration Period (baseline), Day 0 of Treatment Period (last day of Titration Period), Week 12 or end of study visit during the Treatment Period
Population: Safety analysis set (entire study), Full analysis set (treatment period)
Measure: Count of Participants; unit: Participants
Groups:
- Hydrocodone ER (Safety Analysis Set): All enrolled participants who were administered hydrocodone ER tablets at dosages of 15, 30, 45, 60, or 90 mg every 12 hours. Includes days on hydrocodone ER during both the titration and treatment periods.
Arm/Group | Hydrocodone ER (Safety Analysis Set) | Placebo (Double-blind Treatment Period) | Hydrocodone ER (Double-blind Treatment Period)
Number analyzed (Participants) | 623 | 179 | 191
Participants
  >= 1 CS value during study | 29 | 10 | 8
  >= CS value during open-label titration period | 13 | 5 | 2
  >= 1 CS during double-blind treatment period | NA — See values in Hydrocodone ER (Double-blind Treatment Period) column | 8 | 6
  >=CS value at endpoint | NA — See values in Hydrocodone ER (Double-blind Treatment Period) column | 8 | 7

8. Secondary Outcome: Subjective Opiate Withdrawal Scales (SOWS) Total Scores During the Double-Blind Treatment Period
Description: The results of the SOWS were collected in the e-diary daily during the first 4 weeks of the double blind treatment period and then during clinic visits at week 12 or early termination. The SOWS was a self-administered questionnaire used to measure a participant's signs and symptoms of withdrawal from opiates. The scale contained 16 symptoms (such as my nose is running; I feel restless), the participant rated the intensity on a scale of 0 (not at all) to 4 (extremely) for a total score of 0-64. The daily total score for the first 4 weeks was the largest score observed during the time period preceding that visit. For example, the week 1 score for each participant was the largest total score on any day between baseline and the night before the week 1 visit; the week 4 score for each participant was the largest score observed between the week 2 visit and the night before the week 4 visit.
Time Frame: Weeks 1, 2, 4 and Endpoint of the Treatment Period
Population: Full analysis set. Participants contributing to each time point are listed in the time point label.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo (Double-blind Treatment Period) | Hydrocodone ER (Double-blind Treatment Period)
Number analyzed (Participants) | 179 | 191
units on a scale
  Week 1: number analyzed (Participants) | 174 | 186
  Week 1 | 6.9 (7.03) | 6.6 (7.36)
  Week 2: number analyzed (Participants) | 164 | 180
  Week 2 | 5.1 (6.10) | 5.1 (6.89)
  Week 4: number analyzed (Participants) | 151 | 172
  Week 4 | 5.0 (5.52) | 5.5 (6.58)
  Endpoint: number analyzed (Participants) | 176 | 189
  Endpoint | 5.7 (6.70) | 6.1 (7.63)

9. Secondary Outcome: Clinical Opiate Withdrawal Scales (COWS) Total Scores During the Double-Blind Treatment Period
Description: COWS is a clinician-rated scale used to measure a participant's signs and symptoms of withdrawal from opiates, with ratings based only on apparent relationship to withdrawal. The COWS was performed at weeks 1, 2, 4, and 12 (double blind treatment period) or early termination. The scale contained 11 signs/symptoms whose intensity the clinician rated on a scale of 0 to 4 or 5.
  A total score was calculated as the sum of the responses to the 11 signs/symptoms for a total range of 0-48. Withdrawal severity was classified, based on the total score, as follows:
  * 0 to 4=normal
  * 5 to 12=mild
  * 13 to 24=moderate
  * 25 to 36=moderately severe
    * 36=severe
Time Frame: Weeks 1, 2, 4 and Endpoint of the Treatment Period
Population: Full analysis set. Participants contributing to each time point are listed in the time point label.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo (Double-blind Treatment Period) | Hydrocodone ER (Double-blind Treatment Period)
Number analyzed (Participants) | 179 | 191
units on a scale
  Week 1: number analyzed (Participants) | 170 | 181
  Week 1 | 0.9 (1.66) | 0.8 (1.33)
  Week 2: number analyzed (Participants) | 161 | 180
  Week 2 | 0.8 (1.52) | 0.7 (1.13)
  Week 4: number analyzed (Participants) | 149 | 167
  Week 4 | 0.8 (1.33) | 0.6 (1.03)
  Endpoint: number analyzed (Participants) | 174 | 185
  Endpoint | 0.9 (1.49) | 0.7 (1.12)

10. Secondary Outcome: Participants With Potentially Clinically Significant Abnormal Laboratory Values During the Double-Blind Treatment Period
Description: Data represents participants with potentially clinically significant abnormal serum chemistry, hematology and urinalysis values.
  Significance criteria:
  * Blood urea nitrogen: >=10.71 mmol/L
  * Creatinine: >=177 μmol/L
  * Uric acid: M>=625, F>=506 μmol/L
  * Alanine aminotransferase (ALT): >=3* upper limit of normal (ULN)
  * Gamma-glutamyl transpeptidase (GGT): >=3* upper limit of normal (ULN)
  * Serum white blood cells: <=3.0 * 10^9/L
  * Hemoglobin: M<=115, F<=95 g/dL
  * Hematocrit: M<0.37, F<0.32 L/L
  * Eosinophils: >=10.0 %
  * Absolute neutrophils: <=1.0 * 10^9/L
  * Urinalysis: Glucose: >=2 unit increase from baseline
Time Frame: Day 1 up to Week 12 of the Treatment Period
Population: Full analysis set including participants with laboratory assessments. Participants with a postbaseline result for that test are counted in each laboratory tests' label.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Double-blind Treatment Period) | Hydrocodone ER (Double-blind Treatment Period)
Number analyzed (Participants) | 171 | 178
Participants
  Blood urea nitrogen | 3 | 1
  Creatinine | 0 | 1
  Uric acid | 3 | 4
  ALT | 1 | 2
  GGT | 6 | 5
  White blood cells: number analyzed (Participants) | 167 | 171
  White blood cells | 1 | 0
  Hemoglobin: number analyzed (Participants) | 169 | 173
  Hemoglobin | 1 | 2
  Hematocrit: number analyzed (Participants) | 169 | 173
  Hematocrit | 6 | 3
  Eosinophils: number analyzed (Participants) | 167 | 171
  Eosinophils | 1 | 2
  Absolute neutrophils: number analyzed (Participants) | 167 | 171
  Absolute neutrophils | 1 | 2
  Urine glucose: number analyzed (Participants) | 168 | 174
  Urine glucose | 2 | 3

11. Secondary Outcome: Participants With Potentially Clinically Significant Abnormal Vital Sign Values During the Double-Blind Treatment Period
Description: Data represents participants with potentially clinically significant (PCS) vital sign values.
  Significance criteria
  * Pulse - high: >=120 and increase of >= 15 beats/minute from baseline
  * Pulse - low: <=50 and decrease of >=15 beats/minute
  * Systolic blood pressure - high: >=180 and increase >=20 mmHg
  * Systolic blood pressure - low: <=90 and decrease >=20 mmHg
  * Diastolic blood pressure - high: >=105 and increase of >=15 mmHg
  * Diastolic blood pressure - low: <=50 and decrease of >=15 mmHg
Time Frame: Day 1 to Week 12 of the Treatment Period
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Double-blind Treatment Period) | Hydrocodone ER (Double-blind Treatment Period)
Number analyzed (Participants) | 179 | 191
Participants
  Pulse - high | 2 | 1
  Pulse - low | 1 | 1
  Systolic BP - high | 1 | 2
  Systolic BP - low | 2 | 3
  Diastolic BP - high | 0 | 3
  Diastolic BP - low | 0 | 2

12. Secondary Outcome: Participants With Potentially Clinically Significant Abnormal Electrocardiogram Findings During the Double-Blind Treatment Period
Description: Data represents the number of participants with potentially clinically significant (PCS) electrocardiogram findings on the final study visit.
Time Frame: Final study visit (week 12 or end of treatment visit)
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Double-blind Treatment Period) | Hydrocodone ER (Double-blind Treatment Period)
Number analyzed (Participants) | 179 | 191
Participants | 2 | 2

ADVERSE EVENTS:
Time Frame: - Day 1 up to Day 43 (maximum duration) of the Titration Period - Day 1 up to Day 93 (maximum duration) of the Treatment Period
Arm/Group | Hydrocodone ER (Open-Label Titration Period) | Placebo (Double-blind Treatment Period) | Hydrocodone ER (Double-blind Treatment Period)
Serious Adverse Events (participants affected / at risk) | 10/623 | 3/179 | 3/191
Other Adverse Events (participants affected / at risk) | 211/623 | 41/179 | 58/191
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydrocodone ER (Open-Label Titration Period) (N=623) | Placebo (Double-blind Treatment Period) (N=179) | Hydrocodone ER (Double-blind Treatment Period) (N=191)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Tracheal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydrocodone ER (Open-Label Titration Period) (N=623) | Placebo (Double-blind Treatment Period) (N=179) | Hydrocodone ER (Double-blind Treatment Period) (N=191)
Constipation (Gastrointestinal disorders) | 97 (102) | 8 (8) | 27 (29)
Nausea (Gastrointestinal disorders) | 98 (101) | 14 (16) | 20 (23)
Vomiting (Gastrointestinal disorders) | 39 (39) | 6 (6) | 8 (8)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 9 (9) | 8 (9)
Dizziness (Nervous system disorders) | 33 (35) | 4 (4) | 2 (2)
Headache (Nervous system disorders) | 42 (44) | 8 (8) | 11 (11)
Somnolence (Nervous system disorders) | 36 (38) | 2 (2) | 6 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.